CLINICAL TRIAL: NCT02502617
Title: Effect of Intensive Re-nutrition on Eating Disorder Psychopathology, Cognitive Functions, Anxiety, Depression, and Cortisol Level in Severe Anorexia Nervosa
Brief Title: Re-nutrition in Severe Anorexia Nervosa
Acronym: RESAN
Status: Completed | Type: Observational
Sponsor: René Klinkby Støving (Other)
Responsible Party: Sponsor-Investigator, René Klinkby Støving, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: RESAN
Record Dates: First submitted 2015-07-12; First posted 2015-07-20 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Anorexia Nervosa
Keywords: Psychopathology; Cognition; Depression; Nutrition; Cortisol; Anorexia nervosa
MeSH Terms: conditions — Anorexia Nervosa; Depression | interventions — Nutrition Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Weight Improvement: Patients (n = 30) with severe AN, refered to the specialized medical nutrition section at Odense University Hospital are tested three times during nutritional rehabilitation: At admission, at discharge (or drop out) and two-four months after discharge. The first study is carried out not before the third day of hospitalization after acclimatization and water electrolyte correction.
  Interventions: Dietary Supplement: medical nutrition
- Weight-stable: To investigate the re-test effects of the the surveys, outpatients with a stable weight (less than 5%/3 months) with eating disorders (n = 15) are tested twice with 4-6 weeks interval.

INTERVENTIONS:
Dietary Supplement: medical nutrition — The participants are expected to improve their body weight with 10-30% during a closely monitored inpatient-treatment comprising nutritional rehabilitation.
  Groups: Weight Improvement

SUMMARY:
In anorexia nervosa (AN) it still remains to be clarified, which psychiatric symptoms are the direct consequence of malnutrition and adaptation to starvation and which are not. There is clinical consensus that depression/anxiety and cognitive impairments in AN mainly are sequelae to the malnutrition. However, this consensus is largely based on experimental starvation studies of healthy subjects back in 1940s and from famine- and food programs in the third world, whereas evidence from studies on AN is lacking.

The main objective of the study is in the detail to elucidate the short-term changes in the psychopathological profile, depression, anxiety, and cognitive functions in relations to intensive nutritional rehabilitation with weight gain of 10-30% in a specialized medical stabilization unit. Secondarily, it is examined whether cortisol levels are associated with depression/anxiety symptomatology and cognitive impairments. The hypothesis is that an improvement in nutritional status over a short time leads to clinically significant improvements in psychopathology and cognitive functions, which remain 2-3 months after discharge, making the patients more accessible to psychotherapy.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a syndrome characterized by a distorted body image and morbid fear of obesity. Restrictive eating and compensatory behavior in the form of excessive exercising or vomiting result in malnutrition. Repeated revisions of the diagnostic criteria in recent decades have by definition resulted in an increase in prevalence. The disease has the highest mortality among all psychiatric disorders. The majority of deaths is related to malnutrition and its consequences. There is no effective evidence-based treatment. At least 25% remain chronically undernourished and have a long course with prolonged hospitalizations in both psychiatric and medical units, social psychiatric institutions and - support, early retirement and premature death. The etiology remains unknown and it is unclear which of the psychological symptoms that are a consequence of malnutrition, and which ones are premorbid or comorbid.

Depression and anxiety are co-existing and familiar features of patients with AN and can occur in such a degree that it is termed comorbidity. Antidepressant therapy has not shown to have any therapeutic effect of AN. Varying degrees of cognitive impairment are also well known feature of the AN, but in the literature it is only scanty investigated and psychometric analyzed.

In the early stage of the disease, starvation and weight loss can be interpreted as a coping strategy that relieves anxiety and depressive symptoms. If this coping strategy works, then the effect may decreases in line with the severity of malnutrition. There is almost a clinical consensus that depression / anxiety and cognitive impairment in AN is sequelae to malnutrition. But, it is a consensus that rely mainly on experimental studies of healthy subjects back in the postwar years observations from famine and from food programs in the 3rd World. Knowledge of the relationship between psychopathology and malnutrition in AN is still limited to a few and small studies with contradictory conclusions. In a recent study of hospitalized patients, no correlations between body mass index (BMI) and selected psychometric variables could be detected, with the essential limitation that it was a cross-sectional study of a population of patients with a narrow BMI range. To our knowledge, only one longitudinal study on changes in BMI and depressive symptoms have been published. In that study, mean weight gain was a significant predictor of reduced score in several of the "specific" eating disorder symptoms, such as concerns about diet, while weight gain was not a predictor of concern about body nor for depressive symptoms. To our knowledge, no longitudinal re-nutrition studies of the relationship between weight gain and anxiety or cognitive functions has been published.

A consequence of starvation stress is that all the endocrine axes are altered in AN, leading to protein- and energy preserving adaptation. Thus, in particular, increased levels of cortisol is well described in both AN and in patients with primary affective disorders. Depression/anxiety and cognitive impairment is also a well-described side effect of pharmacological treatment with corticosteroids and is well-known symptoms in excess endogenous cortisol production (mb. Cushing). Moreover, neuroanatomical animal studies indicate that cortisol per se has neurotoxic properties and may play a pathogenic role in affective disorders and anxiety. There is preliminary experimental evidence that pharmacological cortisol synthesis inhibition may have therapeutic efficacy in depression. However, so far this is not investigated in AN. In one study, it was found that cortisol levels correlated positively with anxiety and depression.

Center for Eating Disorders at Odense University Hospital is one of three highly specialized national centers in Denmark. Within the center, there is a formalized collaboration between the psychiatric and somatic units. Patients with life-threatening weight loss are primarily hospitalized in the Nutrition section for somatic stabilization and weight gain typically, 10-40%, and then either transferred to the psychiatric department or discharged for two-track psychiatric / somatic outpatient treatment. The Nutrition section receives severely ill patients from the nation. The median BMI of 84 admissions in year 2013 was 13.8 (the range 7.8 - 25.8). Internationally, there are only few somatic units of similar specialization and patient volume, which constitute the basis for studying the effect of intensive re-nutrition per se. The center's organization and patient population is described in several observational and intervention studies.

International and national guidelines recommend that treatment of AN should be interdisciplinary and double-track psychiatric - somatic. But, it is not clear how far and how fast nutritional rehabilitation may have beneficial effects on depression, anxiety and cognitive impairment in patients with severe AN.

ELIGIBILITY:
Inclusion criteria:

- Fulfilling Diagnostic and Statistical Manual (DSM)-5 criteria for AN.

Exclusion Criteria:

* Patients who can not fill Danish-language questionnaires.
* Patients who are primarily hospitalized a few days for water electrolyte correction only.
* Patients with active drug abuse.
* Patients with co-morbid schizophrenia.
* Patients where the psychopharmacological treatment qualitative is changed during the study period.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe AN referred to a specialized unit.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Depression/anxiety and cognitive functions composite outcome measure. | 4-6 months
  Depression/anxiety and cognitive functions composite outcome measure. [Time Frame: 4-6 months] [Safety Issue: No] Admission, discharge, and 2-4 months after discharge. Composite outcome measure consisting of the following psychometry: Beck Depression Inventory version 2 (BDI-II), Hospital Anxiety and Depression Scale (HADS), The Perceived Stress Scale (PSS), Wechsler Memory Scale - Third Edition (WMS-III), Wechsler Adult Intelligent Scale-IV, D2 test, Delis-Kaplan Executive Function System (Trail Making Test, Design Fluency Test and Verbal Fluency Test) and Wisconsin Card Sorting Test - Revised. A total score for each of the psychometric subscales will be calculated and tested in pairs with appropriate corrections for multiple testing.

SECONDARY OUTCOMES:
Eating disorder psychopathology composite outcome measure. | 4-6 months
  Admission, discharge, and 2-4 months after discharge. Composite outcome measure consisting of the following psychometry: Eating Disorder Inventory-3 (EDI-3) and Toronto Alexithymia Scale (TAS-20). A total score for each of the subscales in EDI-3 and for TAS-20 will be calculated and tested in pairs.
Cortisol excretion (nmol Cortisol pr day). | 4-6 months
  Chromatographic mass spectrometric analysis of mixed day urine at admission, discharge, and 2-4 months after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: René K Støving, MD PhD, Principal Investigator — Center for Eating Disorders, Odense University Hospital
Locations (2):
- Denmark (2):
  - Center for Eating Disorders, Department of Endocrinology, Odense University Hospital, Odense
  - René Klinkby Støving, Odense

IPD SHARING:
Plan to Share IPD: No
Data will be entered in Odense Patient data Explorative Network (OPEN).

REFERENCES:
- [Background] Treasure J, Claudino AM, Zucker N. Eating disorders. Lancet. 2010 Feb 13;375(9714):583-93. doi: 10.1016/S0140-6736(09)61748-7. PMID 19931176
- [Background] Pollice C, Kaye WH, Greeno CG, Weltzin TE. Relationship of depression, anxiety, and obsessionality to state of illness in anorexia nervosa. Int J Eat Disord. 1997 May;21(4):367-76. doi: 10.1002/(sici)1098-108x(1997)21:43.0.co;2-w. PMID 9138049
- [Background] Andries A, Gram B, Stoving RK. Effect of dronabinol therapy on physical activity in anorexia nervosa: a randomised, controlled trial. Eat Weight Disord. 2015 Mar;20(1):13-21. doi: 10.1007/s40519-014-0132-5. Epub 2014 Jun 3. PMID 24890912
- [Background] Stoving RK, Andries A, Brixen KT, Bilenberg N, Lichtenstein MB, Horder K. Purging behavior in anorexia nervosa and eating disorder not otherwise specified: a retrospective cohort study. Psychiatry Res. 2012 Jul 30;198(2):253-8. doi: 10.1016/j.psychres.2011.10.009. Epub 2012 Mar 10. PMID 22410588
- [Background] Stoving RK, Andries A, Brixen K, Bilenberg N, Horder K. Gender differences in outcome of eating disorders: a retrospective cohort study. Psychiatry Res. 2011 Apr 30;186(2-3):362-6. doi: 10.1016/j.psychres.2010.08.005. Epub 2010 Sep 9. PMID 20826003
- [Background] Stoving RK, Hangaard J, Hagen C. Update on endocrine disturbances in anorexia nervosa. J Pediatr Endocrinol Metab. 2001 May;14(5):459-80. doi: 10.1515/jpem.2001.14.5.459. PMID 11393567
- [Background] Martins VJ, Toledo Florencio TM, Grillo LP, do Carmo P Franco M, Martins PA, Clemente AP, Santos CD, de Fatima A Vieira M, Sawaya AL. Long-lasting effects of undernutrition. Int J Environ Res Public Health. 2011 Jun;8(6):1817-46. doi: 10.3390/ijerph8061817. Epub 2011 May 26. PMID 21776204
- [Background] Clausen L, Rokkedal K, Rosenvinge JH. Validating the eating disorder inventory (EDI-2) in two Danish samples: a comparison between female eating disorder patients and females from the general population. Eur Eat Disord Rev. 2009 Nov;17(6):462-7. doi: 10.1002/erv.945. PMID 19504471
- [Background] Clausen L, Rosenvinge JH, Friborg O, Rokkedal K. Validating the Eating Disorder Inventory-3 (EDI-3): A Comparison Between 561 Female Eating Disorders Patients and 878 Females from the General Population. J Psychopathol Behav Assess. 2011 Mar;33(1):101-110. doi: 10.1007/s10862-010-9207-4. Epub 2010 Oct 19. PMID 21472023
- [Background] Bagby RM, Taylor GJ, Parker JD. The Twenty-item Toronto Alexithymia Scale--II. Convergent, discriminant, and concurrent validity. J Psychosom Res. 1994 Jan;38(1):33-40. doi: 10.1016/0022-3999(94)90006-x. PMID 8126688
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Beck AT, Steer, R.A., & Brown, G.K. Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation; 1996.
- [Background] Fuss S, Trottier K, Carter J. An investigation of the factor structure of the beck depression inventory-II in anorexia nervosa. Eur Eat Disord Rev. 2015 Jan;23(1):43-50. doi: 10.1002/erv.2338. Epub 2014 Dec 14. PMID 25504530
- [Background] Snaith P, Zigmond AS. Anxiety and depression in general medical settings. BMJ. 1988 Dec 10;297(6662):1544. doi: 10.1136/bmj.297.6662.1544. No abstract available. PMID 3147074
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Garner DM, Olmsted MP, Polivy J, Garfinkel PE. Comparison between weight-preoccupied women and anorexia nervosa. Psychosom Med. 1984 May-Jun;46(3):255-66. doi: 10.1097/00006842-198405000-00007. PMID 6739685
- [Derived] Hemmingsen SD, Lichtenstein MB, Sjogren M, Gudex C, Larsen PV, Stoving RK. Cognitive performance in hospitalized patients with severe or extreme anorexia nervosa. Eat Weight Disord. 2023 Oct 21;28(1):86. doi: 10.1007/s40519-023-01585-w. PMID 37864583
- [Derived] Hemmingsen SD, Jensen NA, Larsen PV, Sjogren JM, Lichtenstein MB, Stoving RK. Cortisol, Depression, and Anxiety Levels Before and After Short-Term Intensive Nutritional Stabilization in Patients With Severe Anorexia Nervosa. Front Psychiatry. 2022 Jul 12;13:939225. doi: 10.3389/fpsyt.2022.939225. eCollection 2022. PMID 35903636
- [Derived] Hemmingsen SD, Lichtenstein MB, Hussain AA, Sjogren JM, Stoving RK. Case report: cognitive performance in an extreme case of anorexia nervosa with a body mass index of 7.7. BMC Psychiatry. 2020 Jun 5;20(1):284. doi: 10.1186/s12888-020-02701-1. PMID 32503476